CLINICAL TRIAL: NCT02706834
Title: A Randomized, Double-Blind (Sponsor-Open), Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Escalating Single Doses of TAK-828 in Healthy Non-Japanese and Japanese Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Escalating Single Doses of TAK-828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-828-1001; U1111-1177-8044 (Registry Identifier: WHO)
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-01

CONDITIONS: Dose Finding Study
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort 1, Sequence I (Experimental): Non-Japanese participants. TAK-828 0.1 mg, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 0.5 mg, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 15 mg, oral solution, fasted, on Day 1 of Period 3; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 1, Sequence II (Experimental): Non-Japanese participants. TAK-828 0.1 mg, oral solution, fasted (after an 8 hour fast) on Day 1 of Period 1; followed by, TAK-828 0.5 mg, oral solution, fasted, on Day 1 of Period 2; followed by, placebo-matching, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 1, Sequence III (Experimental): Non-Japanese participants. TAK-828 0.1 mg, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 15 mg, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 1, Sequence IV (Experimental): Non-Japanese participants. Placebo-matching TAK-828, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 0.5 mg, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 15 mg, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 2, Sequence I (Experimental): Non-Japanese participants. TAK-828 3 mg, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 50 mg, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 200 mg, oral solution, fasted, on Day 1 of Period 3; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 2, Sequence II (Experimental): Non-Japanese participants. TAK-828 3 mg, oral solution, fasted (after an 8 hour fast) on Day 1 of Period 1; followed by, TAK-828 50 mg, oral solution, fasted, on Day 1 of Period 2; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 2, Sequence III (Experimental): Non-Japanese participants. TAK-828 3 mg, oral solution, fasted (after an 8 hour fast) on Day 1 of Period 1; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 200 mg, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 2, Sequence IV (Experimental): Non-Japanese participants. Placebo-matching TAK-828, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 50 mg, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 200 mg, oral solution, fasted, on Day 1 of Period 3; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 4; followed by, TAK-828 100 mg, oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5. There was a 7-day washout period between each period. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 3, Sequence I (Experimental): Japanese participants. TAK-828 15 mg, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 2; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 3. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 3, Sequence II (Experimental): Japanese participants. TAK-828 15 mg, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, placebo-matching TAK-828, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 150 mg, oral solution, fasted, on Day 1 of Period 3. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo
- Cohort 3, Sequence III (Experimental): Japanese participants. Placebo-matching TAK-828, oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1; followed by, TAK-828 100 mg, oral solution, fasted, on Day 1 of Period 2; followed by, TAK-828 150 mg, oral solution, fasted, on Day 1 of Period 3. Each period lasted 4 days with a 7-day washout period between periods.
  Interventions: Drug: TAK-828; Drug: Placebo

INTERVENTIONS:
Drug: TAK-828 — TAK-828 oral solution
Drug: Placebo — TAK-828 placebo-matching oral solution

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single oral doses of TAK-828 in healthy non-Japanese and Japanese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-828. TAK-828 is being tested to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single oral doses of TAK-828 in healthy non-Japanese and Japanese participants.

The study enrolled 36 healthy participants. An interleaving crossover design with placebo substitution was used for Cohorts 1 and 2, and a crossover design was used in Cohort 3. Each cohort consisted of 12 participants, and participants were randomized to treatment sequence to receive TAK-828 or placebo after undergoing a fasting stage of at least 8 hours through intervention periods 1-4 for Cohorts 1 and 2 and through intervention periods 1 - 3 for Cohort 3. The assigned treatment sequence will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need). An additional interventional period 5 (fed state) is planned to be conducted in either cohort 1 or 2, based on the dose of TAK-828 that will be chosen to be studied under fed conditions. Cohorts 1 and 2 were conducted in non-Japanese participants and Cohort 3 in Japanese participants.

This multi-center trial was conducted in the United States. Participants remained confined to the study site from check-in (Day -1) through Day 4 of each intervention period and returned 7 to 10 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria: -

1. Is a healthy male and female (non-child bearing potential) participants.
2. Cohorts 1 and 2: non-Japanese participants aged 18 to 55 years, inclusive, with body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m^ 2), inclusive, and body weight greater than or equal (>=) 50 kilograms (kg).
3. Cohort 3: Japanese participants (born to Japanese parents and grandparents) aged 20 to 55 years, inclusive, with BMI of 18.5 to 25 kg/m^ 2, inclusive, and body weight >= 45 kg.

Exclusion Criteria: -

1. Has used prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to Check-in (Day -1). Herbal supplements and hormone replacement therapy (HRT) must be discontinued 28 days prior to Check-in (Day -1). As an exception, acetaminophen may be used at doses of less than equal to (<=) 1 gram per day (g/day). Limited use of nonprescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-01; Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 01 March 2016 to 17 June 2016.
Pre-assignment Details: Non-Japanese healthy participants were randomized to Cohort 1 or Cohort 2 with 4 different sequences to receive TAK-828 or placebo in a ratio of 9:3. Japanese healthy participants were randomized into Cohort 3 with 3 different sequences to receive TAK-828 or placebo in a ratio of 8:4.
Period: Overall Study
Arm/Group | Cohort 1, Sequence I | Cohort 1, Sequence II | Cohort 1, Sequence III | Cohort 1, Sequence IV | Cohort 2, Sequence I | Cohort 2, Sequence II | Cohort 2, Sequence III | Cohort 2, Sequence IV | Cohort 3, Sequence I | Cohort 3, Sequence II | Cohort 3, Sequence III
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 4
Completed | 1 (Completed = completed study drug) | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 4 | 3 | 3
Not Completed | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Reason Not Specified | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Sequence I | Cohort 1, Sequence II | Cohort 1, Sequence III | Cohort 1, Sequence IV | Cohort 2, Sequence I | Cohort 2, Sequence II | Cohort 2, Sequence III | Cohort 2, Sequence IV | Cohort 3, Sequence I | Cohort 3, Sequence II | Cohort 3, Sequence III | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (10.26) | 29.3 (11.68) | 34.7 (4.16) | 36.7 (9.71) | 28.0 (6.24) | 40.3 (8.39) | 32.3 (10.69) | 40.7 (5.51) | 37.5 (10.02) | 34.3 (6.65) | 43.8 (5.44) | 35.9 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Male | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 4 | 4 | 4 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 2 | 3 | 3 | 3 | 2 | 1 | 3 | 2 | 4 | 4 | 4 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 4 | 4 | 13
  Black or African American | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  White | 2 | 2 | 1 | 2 | 2 | 3 | 3 | 2 | 0 | 0 | 0 | 17
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 36
Height [Mean (Standard Deviation); unit: cm] | 176.3 (3.21) | 176.3 (2.89) | 173.3 (5.69) | 176.7 (1.53) | 169.7 (12.50) | 166.1 (9.54) | 178.0 (4.36) | 170.3 (7.23) | 174.3 (6.24) | 168.5 (5.00) | 173.0 (8.64) | 172.9 (6.82)
Weight [Mean (Standard Deviation); unit: kg] | 81.87 (8.686) | 85.23 (2.686) | 78.60 (9.569) | 83.23 (9.160) | 75.53 (8.173) | 66.87 (8.135) | 81.63 (11.946) | 77.13 (16.354) | 66.73 (1.563) | 65.18 (3.149) | 69.88 (10.806) | 74.93 (10.416)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.28 (1.828) | 27.41 (0.755) | 26.08 (1.765) | 26.65 (2.727) | 26.34 (3.071) | 24.25 (1.772) | 25.73 (3.170) | 26.37 (3.709) | 22.05 (1.864) | 22.96 (0.527) | 23.20 (1.622) | 25.01 (2.584)
Smoking Classification [Number; unit: participants]
  Never Smoked | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 33
  Current Smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Alcohol Classification [Number; unit: participants]
  Never Drunk | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 3 | 2 | 3 | 1 | 16
  Current Drinker | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 11
  Ex-drinker | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 8
  Missing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Xanthine/Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 2 | 4 | 25
  No | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 11
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Surgically Sterile | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Female of Childbearing Potential | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  N/A (Participant is Male) | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 4 | 4 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 up to 30 days after last dose of study drug (up to 85 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: Placebo: Non-Japanese participants in Cohort 1 who received placebo-matching TAK-828 oral solution, fasted (after an 8 hour fast), on Day 1 of Periods 1, 2, 3 or 4.
- Cohort 1: TAK-828 0.1 mg/ Fasted: Non-Japanese participants in Cohort 1 who received TAK-828 0.1 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- Cohort 1: TAK-828 0.5 mg/ Fasted: Non-Japanese participants in Cohort 1 who received TAK-828 0.5 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- Cohort 1: TAK-828 15 mg/ Fasted: Non-Japanese participants in Cohort 1 who received TAK-828 15 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
- Cohort 1: TAK-828 100 mg/ Fasted: Non-Japanese participants in Cohort 1 who received TAK-828 100 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 4.
- Cohort 1: TAK-828 100 mg/ Fed: Non-Japanese participants in Cohort 1 who received TAK-828 100 mg oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5.
- Cohort 2: Placebo: Non-Japanese participants in Cohort 2 who received placebo-matching TAK-828 oral solution, fasted (after an 8 hour fast), on Day 1 of Periods 1, 2, 3 or 4.
- Cohort 2: TAK-828 3 mg/ Fasted: Non-Japanese participants in Cohort 2 who received TAK-828 3 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- Cohort 2: TAK-828 50 mg/ Fasted: Non-Japanese participants in Cohort 2 who received TAK-828 50 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- Cohort 2: TAK-828 200 mg/ Fasted: Non-Japanese participants in Cohort 2 who received TAK-828 200 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
- Cohort 2: TAK-828 100 mg/ Fasted: Non-Japanese participants in Cohort 2 who received TAK-828 100 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 4.
- Cohort 2: TAK-828 100 mg/ Fed: Non-Japanese participants in Cohort 2 who received TAK-828 100 mg oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5.
- Cohort 3: Placebo: Japanese participants in Cohort 3 who received placebo-matching TAK-828 oral solution, fasted (after an 8 hour fast), on Day 1 of Periods 1, 2 or 3.
- Cohort 3: TAK-828 15 mg/ Fasted: Japanese participants in Cohort 3 who received TAK-828 15 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- Cohort 3: TAK-828 100 mg/ Fasted: Japanese participants in Cohort 3 who received TAK-828 100 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- Cohort 3: TAK-828 150 mg/ Fasted: Japanese participants in Cohort 3 who received TAK-828 150 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Number analyzed (Participants) | 10 | 9 | 8 | 7 | 7 | 8 | 9 | 9 | 9 | 9 | 9 | 4 | 12 | 8 | 8 | 6
percentage of participants | 30.0 | 55.6 | 37.5 | 14.3 | 0 | 12.5 | 0 | 11.1 | 11.1 | 11.1 | 22.2 | 0 | 0 | 25.0 | 75.0 | 66.7

2. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-828F (Free Base of TAK-828)
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) Set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma or urine concentration of TAK-828F. Food effect statistical analysis is based on 10 participants who received TAK-828 100 mg under fasted and fed conditions.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- TAK-828 0.1 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 1 who received TAK-828 0.1 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- TAK-828 0.5 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 1 who received TAK-828 0.5 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- TAK-828 3 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 2 who received TAK-828 3 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- TAK-828 15 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 1 who received TAK-828 15 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
- TAK-828 50 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 2 who received TAK-828 50 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- TAK-828 100 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohorts 1 and 2 who received TAK-828 100 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 4.
- TAK-828 100 mg/ Fed in Non-Japanese Participants: Non-Japanese participants in Cohorts 1 and 2 who received TAK-828 100 mg oral solution, fed (high-fat, high-calorie meal 30 minutes prior to administration of study drug), on Day 1 of Period 5.
- TAK-828 200 mg/ Fasted in Non-Japanese Participants: Non-Japanese participants in Cohort 2 who received TAK-828 200 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
- TAK-828 15 mg/ Fasted in Japanese Participants: Japanese participants in Cohort 3 who received TAK-828 15 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 1.
- TAK-828 100 mg/ Fasted in Japanese Participants: Japanese participants in Cohort 3 who received TAK-828 100 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 2.
- TAK-828 150 mg/ Fasted in Japanese Participants: Japanese participants in Cohort 3 who received TAK-828 150 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
Arm/Group | TAK-828 0.1 mg/ Fasted in Non-Japanese Participants | TAK-828 0.5 mg/ Fasted in Non-Japanese Participants | TAK-828 3 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Non-Japanese Participants | TAK-828 50 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fed in Non-Japanese Participants | TAK-828 200 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Japanese Participants | TAK-828 100 mg/ Fasted in Japanese Participants | TAK-828 150 mg/ Fasted in Japanese Participants
Number analyzed (Participants) | 9 | 8 | 9 | 7 | 9 | 16 | 12 | 9 | 8 | 8 | 6
ng/mL | 5.96 (0.982) | 38.6 (3.56) | 247 (28.7) | 1150 (201) | 4820 (1090) | 8900 (1870) | 3730 (850) | 18400 (2950) | 1400 (114) | 9530 (1030) | 14300 (2470)
Statistical Analysis 1: Comparison: TAK-828 100 mg/ Fasted in Non-Japanese Participants vs TAK-828 100 mg/ Fed in Non-Japanese Participants; Food Effect: A linear mixed effect model on the natural log (ln)-transformed parameters was performed with dosing condition as a fixed effect and participant as a random effect using the Kenward-Roger estimation for computing the denominator degrees of freedom. The least squares means and difference of least squared means for the ln-transformed parameters were exponentiated to obtain the geometric means on the original scale; Test type: Non-Inferiority or Equivalence — Bioequivalence interval of 0.80 to 1.25; Point estimate = 0.430, 90% CI 2-sided [0.380 to 0.487] — Exponentiated Least Square Means TAK-828 100 mg Fed/TAK-828 100 mg Fasted

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Time Frame: Day 1 up to 30 days after last dose of study drug (up to 85 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Number analyzed (Participants) | 10 | 9 | 8 | 7 | 7 | 8 | 9 | 9 | 9 | 9 | 9 | 4 | 12 | 8 | 8 | 6
percentage of participants | 0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post-dose
Description: Hematology and Chemistry values that met the following criteria were considered to be markedly abnormal:
  Erythrocytes, Hematocrit and Hemoglobin <0.8*Lower Limit of Normal (LLN) or >1.2*Upper Limit of Normal ULN.; Leukocytes <0.5*LLN or >1.5*ULN; Platelet <75 or >600 10^9/liter (L).
  Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase >3*ULN; Albumin <25 g/L; Bilirubin > 34.2 umol/L; Blood Urea Nitrogen >10.7 mmol/L; Chloride <75 or >126 mmol/L; Creatinine >177 umol/L; Direct Bilirubin >2*ULN; Glucose <2.8 or >19.4 mmol/L; Potassium <3.0 or >6.0 mmol/L; Protein <0.8*LLN or >1.2*ULN; Sodium <130 or >150 mmol/L.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 52 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Number analyzed (Participants) | 10 | 9 | 8 | 7 | 7 | 8 | 9 | 9 | 9 | 9 | 9 | 4 | 12 | 8 | 8 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post-dose
Description: Vital signs measurements that met the following criteria were considered to be markedly abnormal:
  Systolic Blood Pressure (SBP) <85 mmHg or >180 mmHg supine laying face upward) or standing; Diastolic Blood Pressure (DBP) <50 mmHg or >110 mmHg supine or standing; Pulse Rate (PR) <50 beats/minute (bpm) or >120 bpm supine or standing; Temperature <35.6 degrees Celsius (C) or >37.7 degrees C.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 52 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Number analyzed (Participants) | 10 | 9 | 8 | 7 | 7 | 8 | 9 | 9 | 9 | 9 | 9 | 4 | 12 | 8 | 8 | 6
percentage of participants
  SBP <85 mmHg: standing, after 1 minute | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 11.1 | 0 | 8.3 | 0 | 0 | 0
  SBP <85 mmHg: standing, after 3 minutes | 20.0 | 11.1 | 0 | 0 | 0 | 0 | 11.1 | 0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP <50 mmHg: supine, after 5 minutes | 0 | 0 | 0 | 0 | 14.3 | 0 | 0 | 11.1 | 11.1 | 0 | 0 | 0 | 8.3 | 0 | 12.5 | 16.7
  DBP <50 mmHg: standing, after 3 minutes | 10.0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0 | 8.3 | 0 | 12.5 | 16.7
  PR <50 bpm: supine, after 5 minutes | 20.0 | 22.2 | 25.0 | 14.3 | 0 | 25.0 | 33.3 | 22.2 | 22.2 | 22.2 | 22.2 | 50.0 | 0 | 0 | 0 | 16.7
  PR <50 bpm: standing, after 1 minute | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR >120 bpm: standing, after 1 minute | 20.0 | 11.1 | 0 | 0 | 28.6 | 12.5 | 11.1 | 0 | 0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0
  PR <50 bpm: standing, after 3 minutes | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR >120 bpm: standing, after 3 minutes | 20.0 | 11.1 | 25.0 | 0 | 14.3 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: <35.6 C | 10.0 | 22.2 | 0 | 0 | 14.3 | 12.5 | 11.1 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 16.7

6. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) Measurements at Least Once Post-dose
Description: Heart Rate <50 beats per minute (bpm) >120 bpm; QTcB (Bazett's Correction Formula) ≤50 milliseconds (msec) or ≥500 msec OR ≥30 msec change from Baseline and ≥450 msec; QTcF (Fridericia's Correction Formula) ≤50 msec or ≥500 msec OR ≥30 msec change from Baseline (CFB) and ≥450 msec.
Time Frame: Day 1 up to 7 days after last dose of study drug (up to 52 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Number analyzed (Participants) | 10 | 9 | 8 | 7 | 7 | 8 | 9 | 9 | 9 | 9 | 9 | 4 | 12 | 8 | 8 | 6
percentage of participants
  Heart Rate <50 bpm | 20.0 | 33.3 | 25.0 | 28.6 | 0 | 25.0 | 44.4 | 33.3 | 33.3 | 33.3 | 55.6 | 50.0 | 8.3 | 12.5 | 0 | 0
  QTcB: ≥500 msec OR ≥30 msec CFB and ≥450 msec | 0 | 0 | 0 | 0 | 0 | 25.0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 12.5 | 0

7. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-828F (Free Base of TAK-828)
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) Set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma or urine concentration of TAK-828F.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | TAK-828 0.1 mg/ Fasted in Non-Japanese Participants | TAK-828 0.5 mg/ Fasted in Non-Japanese Participants | TAK-828 3 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Non-Japanese Participants | TAK-828 50 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fed in Non-Japanese Participants | TAK-828 200 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Japanese Participants | TAK-828 100 mg/ Fasted in Japanese Participants | TAK-828 150 mg/ Fasted in Japanese Participants
Number analyzed (Participants) | 9 | 8 | 9 | 7 | 9 | 16 | 12 | 9 | 8 | 8 | 6
hours (h) | 1.00 [0.500 to 1.13] | 1.00 [0.517 to 2.00] | 1.00 [0.500 to 1.00] | 1.00 [1.00 to 1.50] | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 1.02] | 3.50 [1.00 to 4.00] | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 2.00] | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 1.03]

8. Secondary Outcome: t1/2z: Terminal Disposition Phase Half-Life for TAK-828F (Free Base of TAK-828)
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) Set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma or urine concentration of TAK-828F. T1/2z was not calculated for the TAK-828 0.1 mg arm because Lambda z, required for the calculation, was not calculated due to the lack of a well-defined terminal elimination phase.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TAK-828 0.1 mg/ Fasted in Non-Japanese Participants | TAK-828 0.5 mg/ Fasted in Non-Japanese Participants | TAK-828 3 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Non-Japanese Participants | TAK-828 50 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fed in Non-Japanese Participants | TAK-828 200 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Japanese Participants | TAK-828 100 mg/ Fasted in Japanese Participants | TAK-828 150 mg/ Fasted in Japanese Participants
Number analyzed (Participants) | 0 | 7 | 9 | 7 | 9 | 16 | 12 | 9 | 8 | 8 | 6
h |  | 5.38 (0.568) | 4.94 (1.11) | 6.53 (1.14) | 7.51 (1.95) | 7.53 (1.32) | 7.04 (0.701) | 7.97 (1.42) | 6.71 (1.37) | 6.71 (0.950) | 6.44 (0.406)

9. Secondary Outcome: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity Calculated Using the Observed Value of the Last Quantifiable Concentration for TAK-828F (Free Base of TAK-828)
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 72 hours) post-dose
Population: PK Set included participants who received at least 1 dose of study drug and had at least 1 measurable plasma or urine concentration of TAK-828F.Food effect statistical analysis is based on 10 participants who received TAK-828 100 mg fasted and fed.AUC∞ was not calculated for TAK-828 0.1 mg arm due to lack of well-defined terminal elimination phase.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TAK-828 0.1 mg/ Fasted in Non-Japanese Participants | TAK-828 0.5 mg/ Fasted in Non-Japanese Participants | TAK-828 3 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Non-Japanese Participants | TAK-828 50 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fasted in Non-Japanese Participants | TAK-828 100 mg/ Fed in Non-Japanese Participants | TAK-828 200 mg/ Fasted in Non-Japanese Participants | TAK-828 15 mg/ Fasted in Japanese Participants | TAK-828 100 mg/ Fasted in Japanese Participants | TAK-828 150 mg/ Fasted in Japanese Participants
Number analyzed (Participants) | 0 | 7 | 9 | 7 | 9 | 16 | 12 | 9 | 8 | 8 | 6
ng*h/mL |  | 214 (30.4) | 1150 (211) | 5930 (1430) | 23100 (5400) | 45400 (10300) | 38000 (7370) | 106000 (20800) | 8560 (1610) | 54600 (13400) | 83700 (16400)
Statistical Analysis 1: Comparison: TAK-828 100 mg/ Fasted in Non-Japanese Participants vs TAK-828 100 mg/ Fed in Non-Japanese Participants; Food Effect: A linear mixed effect model on the natural log (ln)-transformed parameters was performed with dosing condition as a fixed effect and participant as a random effect using the Kenward-Roger estimation for computing the denominator degrees of freedom. The least squares means and difference of least squared means for the ln-transformed parameters were exponentiated to obtain the geometric means and ratios of geometric means on the original scale; Test type: Non-Inferiority or Equivalence — Bioequivalence interval of 0.80 to 1.25; Point estimate = 0.896, 90% CI 2-sided [0.833 to 0.964] — Exponentiated Least Square Means TAK-828 100 mg Fed/TAK-828 100 mg Fasted

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days after last dose of study drug (up to 85 days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Cohort 2: TAK-828 200 mg/ Fasted: Cohort 2: TAK-828 200 mg/ Fasted Non-Japanese participants in Cohort 2 who received TAK-828 200 mg oral solution, fasted (after an 8 hour fast), on Day 1 of Period 3.
Arm/Group | Cohort 1: Placebo | Cohort 1: TAK-828 0.1 mg/ Fasted | Cohort 1: TAK-828 0.5 mg/ Fasted | Cohort 1: TAK-828 15 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fasted | Cohort 1: TAK-828 100 mg/ Fed | Cohort 2: Placebo | Cohort 2: TAK-828 3 mg/ Fasted | Cohort 2: TAK-828 50 mg/ Fasted | Cohort 2: TAK-828 200 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fasted | Cohort 2: TAK-828 100 mg/ Fed | Cohort 3: Placebo | Cohort 3: TAK-828 15 mg/ Fasted | Cohort 3: TAK-828 100 mg/ Fasted | Cohort 3: TAK-828 150 mg/ Fasted
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9 | 0/8 | 0/7 | 0/7 | 0/8 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/4 | 0/12 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 5/9 | 3/8 | 1/7 | 0/7 | 1/8 | 0/9 | 1/9 | 1/9 | 1/9 | 2/9 | 0/4 | 0/12 | 2/8 | 6/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=10) | Cohort 1: TAK-828 0.1 mg/ Fasted (N=9) | Cohort 1: TAK-828 0.5 mg/ Fasted (N=8) | Cohort 1: TAK-828 15 mg/ Fasted (N=7) | Cohort 1: TAK-828 100 mg/ Fasted (N=7) | Cohort 1: TAK-828 100 mg/ Fed (N=8) | Cohort 2: Placebo (N=9) | Cohort 2: TAK-828 3 mg/ Fasted (N=9) | Cohort 2: TAK-828 50 mg/ Fasted (N=9) | Cohort 2: TAK-828 200 mg/ Fasted (N=9) | Cohort 2: TAK-828 100 mg/ Fasted (N=9) | Cohort 2: TAK-828 100 mg/ Fed (N=4) | Cohort 3: Placebo (N=12) | Cohort 3: TAK-828 15 mg/ Fasted (N=8) | Cohort 3: TAK-828 100 mg/ Fasted (N=8) | Cohort 3: TAK-828 150 mg/ Fasted (N=6)
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=10) | Cohort 1: TAK-828 0.1 mg/ Fasted (N=9) | Cohort 1: TAK-828 0.5 mg/ Fasted (N=8) | Cohort 1: TAK-828 15 mg/ Fasted (N=7) | Cohort 1: TAK-828 100 mg/ Fasted (N=7) | Cohort 1: TAK-828 100 mg/ Fed (N=8) | Cohort 2: Placebo (N=9) | Cohort 2: TAK-828 3 mg/ Fasted (N=9) | Cohort 2: TAK-828 50 mg/ Fasted (N=9) | Cohort 2: TAK-828 200 mg/ Fasted (N=9) | Cohort 2: TAK-828 100 mg/ Fasted (N=9) | Cohort 2: TAK-828 100 mg/ Fed (N=4) | Cohort 3: Placebo (N=12) | Cohort 3: TAK-828 15 mg/ Fasted (N=8) | Cohort 3: TAK-828 100 mg/ Fasted (N=8) | Cohort 3: TAK-828 150 mg/ Fasted (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Foreign body reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Per an audit performed at the study site that enrolled Cohort 3, noncompliance to Good Clinical Practice (GCP) was identified and prevented confirmed reliability of the data collected. Data was still analyzed and results are reported in this posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.